CLINICAL TRIAL: NCT06442475
Title: Low Dose Mosunetuzumab for Indolent B-Cell Lymphoma
Brief Title: Low Dose Mosunetuzumab for the Treatment of Patients With Indolent B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124175; NCI-2024-02289 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20417 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Ann Arbor Stage II Follicular Lymphoma; Ann Arbor Stage II Marginal Zone Lymphoma; Ann Arbor Stage III Follicular Lymphoma; Ann Arbor Stage III Marginal Zone Lymphoma; Ann Arbor Stage IV Follicular Lymphoma; Ann Arbor Stage IV Marginal Zone Lymphoma; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (mosunetuzumab) (Experimental): Patients receive mosunetuzumab IV over 2-4 hours on days 1, 8, 15 and 22. Patients also undergo blood sample collection and PET/CT on study. Patients may undergo CT and/or MRI as clinically indicated and may undergo collection of oral and/or rectal swabs on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Mosunetuzumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood, oral, and/or rectal sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Mosunetuzumab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT 4465A; BTCT-4465A; BTCT4465A; CD20/CD3 BiMAb BTCT4465A; Lunsumio; Mosunetuzumab-axgb; RG 7828; RG-7828; RG7828; RO7030816
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests the safety, side effects and effectiveness of mosunetuzumab in treating patients with slow growing (indolent) B-cell lymphoma. Mosunetuzumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive mosunetuzumab intravenously (IV) over 2-4 hours on days 1, 8, 15 and 22. Patients also undergo blood sample collection and positron emission tomography (PET)/computed tomography (CT) on study. Patients may undergo CT and/or magnetic resonance imaging (MRI) as clinically indicated and may undergo collection of oral and/or rectal swabs on study.

After completion of study treatment, patients are followed up at week 13, at 6 months, and then for up to 5 years per institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at time of signing informed consent
* Capable of understanding and providing written informed consent
* Histologically confirmed indolent B-cell non-Hodgkin lymphoma with no prior therapy for lymphoma. (Prior peptide-based therapeutic vaccines are allowed.) Eligible histologies include:

  * Follicular lymphoma (grade 1-2 or 3A)
  * Marginal zone lymphoma
* Ann Arbor stage II-IV disease
* No prior therapy for lymphoma
* Have low-tumor burden disease, defined by Groupe D'Etude des Lymphomes Folliculaires (GELF) criteria:

  * Nodal or extranodal tumor mass < 7 cm
  * Involvement of less than 3 nodal sites with a diameter > 3 cm
  * No systemic or B symptoms
  * No splenomegaly > 16 cm by imaging
  * No local risk of vital organ compression
  * No pleural or peritoneal serous effusions
  * No leukemic phase (> 5,0000/ uL circulating lymphocytes)
  * No significant cytopenias defined as platelets < 100,000/uL, hemoglobin < 10 g/dL, or absolute neutrophil count (ANC) < 1500/ uL
* Have measurable nodal disease, including at least 1 disease site measuring at least 1.5 cm in longest dimension on CT or fludeoxyglucose F-18 (FDG)-PET, or a FDG-avid extranodal measurable site measuring at least 1.0 cm in longest dimension. Measurable disease also includes spleen size more than 13 cm in vertical length
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Creatinine clearance ≥ 50 mL/min calculated by Cockcroft-Gault equation
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN), except in patients with Gilbert's syndrome who may have a total bilirubin up to ≤ 3 x ULN
* Aspartate aminotransferase (AST) ≤ 3 x the ULN
* Alanine aminotransferase (ALT) ≤ 3 x the ULN
* Gamma glutamyl transferase (GGT) ≤ 3 x the ULN
* Negative serum or urine pregnancy test within 7 days of initiating mosunetuzumab for women of childbearing potential, defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year
* Fertile male and woman of childbearing potential must agree to use highly effective contraceptive methods from start of treatment to at least 3 months after the last dose of mosunetuzumab

Exclusion Criteria:

* History of severe allergic reaction to monoclonal antibody therapy
* History of a second primary malignancy that could affect compliance with the protocol or interpretation of results except with permission of the principal investigator. Malignancies treated curatively or at low-risk of progressing at the judgment of the principal investigator (PI) may be included
* Known active and uncontrolled bacterial, viral, fungal, mycobacterial, or other infection at study enrollment
* Infection with human immunodeficiency virus (unless viral load is undetectable and CD4 count ≥ 200)
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HbBsAg] serology):

  * Patients with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable at the time of screening. These patients must be willing to undergo monthly DNA testing and appropriate antiviral therapy as indicated by institutional standards
* Autoimmune disease requiring active therapy
* History of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* Evidence of significant concurrent disease or medical condition that could interfere with the conduct of the study, or put the patient at significant risk including, but not limited to, significant cardiovascular disease (e.g., New York Heart Association class III or IV cardiac disease, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Ongoing systemic corticosteroid treatment, with the exception of corticosteroid use for other (non-tumor and non-immunosuppressive) indications up to a maximum of 10 mg/day of prednisone or equivalent
* Prior use of any monoclonal antibody within 4 weeks before the first mosunetuzumab administration
* Prior solid organ transplantation
* Pregnant or breast-feeding women, or intending to become pregnant during the study or within 3 months of the last dose of mosunetuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Overall response (OR) | Up to week 13
  OR will be defined as complete response and partial response at the end of therapy based on the latest version of Lugano criteria. Response rates will be calculated using simple binomial proportions and the corresponding 95% confidence interval will be derived.

SECONDARY OUTCOMES:
Incidence of adverse events (AE's) | Up to 30 days after last dose of study treatment
  All AEs will be graded in severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. AEs will be summarized by type, severity, duration, and attribution.
Incidence of grade 3 or greater cytokine release syndrome (CRS) | Up to 30 days after last dose of study treatment
  CRS will be graded by the American Society for Transplantation and Cellular Therapy Consensus Grading system.
Incidence of Immune Effector Cell Associated Neurotoxicity syndrome | Up to 30 days after last dose of study treatment
Progression free survival (PFS) | At initiation of study treatment to disease progression, up to 5 years
  Kaplan-Meier methodology will be used to estimate PFS.
Duration of response | Up to 5 years
Time to next lymphoma treatment | At initiation of study treatment to initiation of next therapy, up to 5 years
  Kaplan-Meier methodology will be used to estimate time to next lymphoma treatment.
Time to cytotoxic treatment | At initiation of study treatment to initiation of cytotoxic treatment, up to 5 years
  Kaplan-Meier methodology will be used to estimate time to cytotoxic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No